CLINICAL TRIAL: NCT05501730
Title: Utilization of the Quantra QPlus System to Guide the Management of Blood Product Transfusions in Cardiac Surgery Patients: Effects on Clinical and Economic Outcomes
Brief Title: Use of the Quantra QPlus Sytem in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-038
Record Dates: First submitted 2022-07-26; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac surgery; Quantra; Viscoelastic testing; Coagulation; QPlus
MeSH Terms: conditions — Cardiovascular Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pre-Quantra: Patients undergoing cardiac surgery prior to the introduction of the Quantra.
- Post-Quantra: Patients undergoing cardiac surgery after the introduction of the Quantra.
  Interventions: Diagnostic Test: Quantra QPlus System

INTERVENTIONS:
Diagnostic Test: Quantra QPlus System — Coagulation monitoring system
  Groups: Post-Quantra

SUMMARY:
Single center retrospective study evaluating the impact of using the Quantra QPlus System to guide transfusion decisions on postoperative outcomes in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Yavapai Regional Medical Center (YRMC) implemented the Quantra QPlus System to aid in their efforts to effectively reduce the transfusion rate of allogenic blood products and improve outcomes in patients undergoing cardiac surgery. Use of the Quantra to guide decisions related to the use of blood products in cardiac surgery patients began in 2019. In this retrospective study, YRMC evaluated the impact of using the Quantra QPlus System to guide transfusion decisions on postoperative outcomes in patients undergoing cardiac surgery.

ELIGIBILITY:
* Pre-Quantra Group: All consecutive patients undergoing cardiac surgical procedures during the period from January 2019 to September 2019 (n=64)
* Post-Quantra Group: All consecutive patients undergoing cardiac surgical procedures during the period from May 2020 to April 2021 (n=64)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery performed by the same surgical team.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Blood product utilization | Intraoperative - during surgery
  Units of blood products administered to patient
Blood product utilization | Postoperative - after surgery throughout the rest of the hospital stay, assessed up to 30 days
  Units of blood products administered to patient
Cost of blood products | Throughout the entire hospital stay, assessed up to 30 days
  Total cost of blood products administered to patient

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tibi, MD, Principal Investigator — Yavapai Regional Medical Center
Locations (1):
- Yavapai Regional Medical Center, Prescott, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tibi P, Thompson J, Attaran S, Black E. Retrospective study assessing outcomes in cardiac surgery after implementation of Quantra. J Cardiothorac Surg. 2023 Apr 17;18(1):149. doi: 10.1186/s13019-023-02245-x. PMID 37069685